CLINICAL TRIAL: NCT00390988
Title: Comparison of Capillary and Venous Blood Count Parameters
Brief Title: Capillary and Venous Blood Count Parameters
Status: Completed | Type: Observational
Sponsor: University of Magdeburg (Other)
Other Study IDs: MD FME 45/06
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Hematological Diseases; Healthy Volunteers
Keywords: blood count; capillary; venous; Adult; reference values
MeSH Terms: conditions — Hematologic Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: blood sampling

SUMMARY:
The purpose of this study is to compare capillary blood count parameters with the corresponding venous samples to verify the hypothesis that capillary and venous blood count parameters are equivalent.

DETAILED DESCRIPTION:
In patients with haematological diseases regular blood count analyses are necessary. In haematology, capillary blood count analyses became established in routine diagnostics. The method and procedure of capillary blood sampling is well accepted by both the patients and the medical personal for a long time. However, only venous values are generally accepted in clinical routine. It is important to know whether or how capillary blood gives discrepant results for the various parameters. Values for therapeutic decisions, e.g. transfusion, are only known for venous values. So far, there are only deficient data available. Therefore, the aim of this study is (i) to compare capillary blood count parameters with the corresponding venous samples to verify the hypothesis that capillary and venous blood count parameters are equivalent, (ii) to include an adequate large number of adult haematological patients (with low and high values) and healthy adults, (iii) to obtain difference values for conversation of measured capillary values into the corresponding venous values.

ELIGIBILITY:
Inclusion Criteria:

* Patients with haematological diseases ≥18 years
* Healthy volunteers ≥18 years
* Informed consent
* No participation in another study 3 month before and during the study

Exclusion Criteria:

* Subjects <18 years
* Healthy subjects with acute or chronic infections and autoimmune or malignant diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Jentsch-Ullrich, Dr., Principal Investigator — University Hospial Magdeburg, Division of Haematoloy/Oncology, Leipziger Str. 44, D-39120 Magdeburg, Germany

REFERENCES:
- [Result] Schalk E, Heim MU, Koenigsmann M, Jentsch-Ullrich K. Use of capillary blood count parameters in adults. Vox Sang. 2007 Nov;93(4):348-53. doi: 10.1111/j.1423-0410.2007.00978.x. PMID 18070280
- [Result] Schalk E, Scheinpflug K, Mohren M. Correlation of capillary and venous absolute neutrophil counts in adult hematological patients and normal controls. Am J Hematol. 2008 Jul;83(7):605. doi: 10.1002/ajh.21163. No abstract available. PMID 18306364